CLINICAL TRIAL: NCT04979481
Title: We R Native: Designing and Evaluating Technologies to Promote Adolescent Mental Health
Brief Title: BRAVE Study: Designing and Evaluating Technologies to Promote Adolescent Mental Health
Acronym: BRAVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwest Portland Area Indian Health Board (Other)
Collaborators: mHealth Impact Lab (Unknown)
Responsible Party: Principal Investigator, Stephanie Craig Rushing, Project Director, Northwest Portland Area Indian Health Board
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 1384639
Record Dates: First submitted 2021-07-14; First posted 2021-07-28 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Mental Health Wellness 1
Keywords: adolescent
MeSH Terms: interventions — Microscopy, Electron, Scanning Transmission

STUDY DESIGN:
Intervention Model Description: Teens and young adults enrolled in the study received either: 8 weeks of BRAVE text messages or 8 weeks of STEM text messages; and then crossed over to the other arm and received the next set of messages.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BRAVE Intervention Arm (Experimental): The BRAVE campaign included 3-5 text messages per week, including 1 role model video per week and a related image.
  Interventions: Behavioral: BRAVE
- STEM Control Arm (Active Comparator): The STEM campaign included 3-5 text messages per week for 8 weeks, including 1 role model video per week and a related image.
  Interventions: Behavioral: STEM

INTERVENTIONS:
Behavioral: BRAVE — The BRAVE campaign included 3-5 text messages per week for 8 weeks, including 1 role model video per week and a related image. The role model videos (1-3 minutes each) featured relatable characters experiencing and addressing violent behavior, alcohol misuse, and suicidality (through the eyes of a perpetrator, an intimate partner violence survivor, and a peer bystander), intended to demonstrated important coping and help-seeking skills.
  Arms: BRAVE Intervention Arm
Behavioral: STEM — The STEM campaign included 3-5 text messages per week for 8 weeks, including 1 role model video per week and a related image. The series promoted STEM career pathways and highlighted Native professionals in Science, Technology, Engineering, Math, and Medical careers.
  Arms: STEM Control Arm

SUMMARY:
The BRAVE study is a randomized controlled trial carried out by the Northwest Portland Area Indian Health Board and the mHealth Impact Lab. The team recruited 2,330 AI/AN teens and young adults nationwide (15-24 years old) via social media channels and text message and enrolled 1,030 to participate in the 9-month study. Teens and young adults enrolled in the study received either: 8 weeks of BRAVE text messages designed to improve mental health, help-seeking skills, and promote cultural pride and resilience; or 8 weeks of Science Technology Engineering and Math (STEM) text messages, designed to elevate and re-affirm Native voices in science, technology, engineering, math and medicine; and then received the other set of messages. Retention in the study was high, with 87% of participants completing both BRAVE and STEM intervention arms.

DETAILED DESCRIPTION:
There are approximately 2.1 million self-identified American Indian and Alaska Native (AI/AN or Native) youth under the age of 24 living in the United States. Like many teens, AI/AN youth report frequent technology use and poor mental health outcomes, including trauma, stress, anxiety, depression, and suicidality.

To support Native youth, the Northwest Portland Area Indian Health Board (NPAIHB) launched We R Native in 2012, a holistic health resource for Native youth, by Native youth (www.weRnative.org).

While this broad reach and utilization is promising, more focused research is needed to better understand the acceptability and usability of the mental health messages delivered by We R Native, and systematic research is needed to determine whether We R Native's messages actually improve mental health and resilience, teach mental health skills (like coping skills, mindfulness, help-seeking, and use of suicide prevention chat-lines, etc.), and promote healthy social norms - all protective factors against suicide and substance abuse.

Housed at the Colorado School of Public Health, the mission of the mHealth Impact Lab is to facilitate the rapid and rigorous development, implementation, and evaluation of mobile and digital technology for health promotion and disease prevention that address inequalities in health outcomes.

The research teams tested whether We R Native's BRAVE messages improved self-efficacy and behaviors related to mental health, resilience, and cultural pride; as well as the relative impact of user engagement.

The BRAVE study will improve the relevance, efficacy, and utilization of mental health resources delivered through We R Native' messaging channels - reaching a high-risk, underserved population - and will create new mechanisms to monitor and evaluate the impact of mHealth interventions. Both teams are committed to sharing resultant data collection tools and processes with those working in the field.

ELIGIBILITY:
Inclusion Criteria:

* The study included self-identified American Indian and Alaska Native youth
* Age 15-24 years old

Exclusion Criteria:

-Participants were required to have a cell phone with text message capabilities

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1030 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Health | Up to 8 months
  Changes in mean scores of perceived mental, physical, and spiritual health
Resilience | Up to 8 months
  Proportion of respondents that report higher mean scores on resilience
Positive Coping | Up to 8 months
  Proportion of respondents that report higher mean scores of coping skills
Self-esteem | Up to 8 months
  Proportion of respondents who report higher mean scores of self-satisfaction, having good qualities, pride, self-worth, and self-respect

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Craig Rushing, PhD, Principal Investigator — Principal Investigator
Locations (1):
- NPAIHB, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan in place at this time.

REFERENCES:
- [Background] Craig Rushing S, Kelley A, Hafner S, Stephens D, Singer M, Bingham D, Caughlan C, Fatupaito B, Gaston A, Ghost Dog T, Smith P, Love Brown D, McCray C. The BRAVE Study: Formative Research to Design a Multimedia Intervention for American Indian and Alaska Native Young Adults. Am Indian Alsk Native Ment Health Res. 2021;28(1):71-102. doi: 10.5820/aian.2801.2021.71. PMID 33844480
- [Result] Stephens D, Peterson R, Singer M, Johnson J, Rushing SC, Kelley A. Recruiting and Engaging American Indian and Alaska Native Teens and Young Adults in a SMS Help-Seeking Intervention: Lessons Learned from the BRAVE Study. Int J Environ Res Public Health. 2020 Dec 16;17(24):9437. doi: 10.3390/ijerph17249437. PMID 33339260
- [Derived] Wrobel J, Silvasstar J, Peterson R, Sumbundu K, Kelley A, Stephens D, Craig Rushing S, Bull S. Text Messaging Intervention for Mental Wellness in American Indian and Alaska Native Teens and Young Adults (BRAVE Study): Analysis of User Engagement Patterns. JMIR Form Res. 2022 Feb 25;6(2):e32138. doi: 10.2196/32138. PMID 35212633
- [Derived] Craig Rushing S, Kelley A, Bull S, Stephens D, Wrobel J, Silvasstar J, Peterson R, Begay C, Ghost Dog T, McCray C, Love Brown D, Thomas M, Caughlan C, Singer M, Smith P, Sumbundu K. Efficacy of an mHealth Intervention (BRAVE) to Promote Mental Wellness for American Indian and Alaska Native Teenagers and Young Adults: Randomized Controlled Trial. JMIR Ment Health. 2021 Sep 15;8(9):e26158. doi: 10.2196/26158. PMID 34524092